CLINICAL TRIAL: NCT00250588
Title: Reducing Barriers to Care for Vulnerable Children With Asthma
Brief Title: Problem-Solving Skills Training to Improve Care for Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R40 MC 00331
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: Asthma; Child; Problem-solving; Quality of Life; Barriers to Care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Problem solving + care coordination (Experimental): Problem solving skills training and asthma care coordination
  Interventions: Behavioral: Problem solving skills training; Behavioral: Asthma care coordination; Other: Usual Care
- Asthma care coordination (Experimental): Asthma care coordination
  Interventions: Behavioral: Asthma care coordination; Other: Usual Care
- Wait-list control (Active Comparator): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Problem solving skills training — See description in Results
  Arms: Problem solving + care coordination
Behavioral: Asthma care coordination — See description in Results
  Arms: Asthma care coordination; Problem solving + care coordination
Other: Usual Care — Usual clinical care

SUMMARY:
The purpose of this study is to determine whether Problem-Solving Skills Training is effective in reducing barriers to health care and improving health-related quality of life for children with persistent asthma.

DETAILED DESCRIPTION:
Brief description: This 4-year research project will develop and test culturally and linguistically appropriate brief interventions to reduce barriers to health care for vulnerable children with persistent asthma.

Background: The U.S. health system presents formidable challenges to the timely receipt of high quality care, especially for vulnerable children (e.g., those in families of color, lower SES, limited English ability). This population is at greatest risk for poor health outcomes. Children with asthma are an important vulnerable subgroup. Asthma, with an estimated prevalence of 6.9%, is the most common chronic condition in children. It is the most frequent reason for pediatric hospitalization and is a condition with documented disparities in care outcomes.

A promising strategy for overcoming the barriers to quality care that these children encounter is the use of care coordinators who educate parents and children, connect the family with needed resources, and coordinate care from different settings. Care coordination has been shown effective in improving receipt of appropriate asthma services and health outcomes for children with asthma. Despite this evidence, there is concern that the effects of care coordination may not be maintained once these services end. This is particularly important given financial pressures to reduce the length and intensity of such services. In order to maintain the gains achieved during care coordination, families need to be able to identify and overcome barriers to care for and by themselves. This can be achieved through the use of Problem Solving Therapy, a documented behavioral method for teaching families the skills they need to resolve daily problems and improve adherence to medical regimens for children with chronic health conditions.

Study Goals: The overall goal of this project is to improve the quality of care and health outcomes for vulnerable children with asthma. The specific aims of this two-phase project are:

* (Phase I) to adapt, in collaboration with community health workers and parents, existing materials to create two culturally and linguistically appropriate treatment manuals: a Care Coordination Treatment Manual that will standardize the delivery of culturally and linguistically appropriate home-based care coordination and asthma-specific education, and a Problem Solving Therapy Treatment Manual tailored to asthma that will include a detailed, step-by-step guide for implementing this approach to reduce barriers to care.
* (Phase II) to use the manuals developed in Phase I to perform a randomized controlled clinical trial to evaluate the effectiveness of two brief interventions involving Care Coordination and tailored Problem Solving Therapy (tPST) in improving and maintaining improvement in health care quality and health-related quality of life for children with asthma.

Evidence for the efficacy of tPST and the availability of culturally and linguistically appropriate treatment manuals should spur diffusion of this innovation to other practitioners and programs seeking evidence-based, optimal clinical management strategies.

Methodology:

Phase I. Existing materials for the Care Coordination and tPST manuals will be edited and/or rewritten to make them specific to asthma. Then both the manuals and the proposed interventions will be assessed for cultural acceptability though two series of parallel focus groups: one for parents of children with asthma, and the other for home visitors already providing care coordination for families of children with asthma. The revised educational materials will then be translated into Spanish.

Phase II. Children ages 2-12 years with persistent asthma and their families (n = 366) will be randomized into two brief interventions:

1. tPST (six sessions) plus Care Coordination (six home visits over 3 months) versus a Wait List control group (usual care) to evaluate the intervention's effectiveness in improving outcomes 3 months after baseline.
2. tPST versus Care Coordination and Wait List to evaluate the intervention's effectiveness in maintaining outcomes 9 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Child age 2 to 12 years old, inclusive
* Diagnosis of persistent asthma (mild, moderate, or severe) according to NHLBI criteria
* Family speaks English or Spanish

Exclusion Criteria:

* Family does not speak English or Spanish
* Child has other comorbid conditions that would affect care or outcomes

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2003-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seid, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Seid M, Varni JW, Gidwani P, Gelhard LR, Slymen DJ. Problem-solving skills training for vulnerable families of children with persistent asthma: report of a randomized trial on health-related quality of life outcomes. J Pediatr Psychol. 2010 Nov;35(10):1133-43. doi: 10.1093/jpepsy/jsp133. Epub 2010 Jan 8. PMID 20061311
- [Derived] Seid M. Barriers to care and primary care for vulnerable children with asthma. Pediatrics. 2008 Nov;122(5):994-1002. doi: 10.1542/peds.2007-3114. PMID 18977978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 11, 2004 and January 15, 2007. The final T3 follow up was completed on October 16, 2007.
Groups:
- Care Coordination: The 5-session (45-60 minutes, weekly) CC was based on NHLBI guidelines and the RWJF's Allies Against Asthma community health worker model (Friedman et al., 2006) and was delivered by two bachelor's level bilingual, bicultural asthma home visitors. The home visitors implemented a structured set of educational interventions, with written materials in English or Spanish, on the following topics: what is asthma, asthma medications and devices, asthma action plan, how to recognize and respond to symptom onset, and how to reduce irritants and allergens in the home. Home visitors referred families, when necessary, to existing health insurance enrollment assistance, smoking cessation, and other community support services. Home visitors communicated with the primary care provider via FAX, giving summaries of interventions, updates on progress, and noting family difficulties and needs (for example, needing equipment, prescriptions, or an (updated) asthma treatment plan).
- Care Coordination+Problem Solving: The CC+PST consisted of CC plus a 6-session (45-60 minutes, weekly) problem-solving skills training intervention. Participants are taught to approach problems proactively, define the problem, generate alternative solutions, choose the best, implement the solution, and evaluate how well that solution worked. Session 1 was devoted to rapport building, understanding the relevant social and medical situation, presenting an overview of the PST curriculum, and assigning the first homework - identifying a solvable problem. Session 2 reviewed prior homework, introduced the idea of developing alternative solutions, and assigned homework - defining and evaluating options. Session 3 reviewed homework, developed an action plan and assigned homework - implementing the action plan. Sessions 4-6 depended on the outcome of the actions, focusing on alternative plans if the results of the action plan were not satisfactory to the client or on additional problems if the results were satisfactory.
- Standard Care: The standard care wait list control group received ongoing asthma care from their place of care during the trial. They were offered the CC+PST intervention after the T3 follow up.
Period: Overall Study
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care
Started | 81 | 84 | 87
Completed | 72 | 65 | 74
Not Completed | 9 | 19 | 13
Not completed — Withdrawal by Subject | 3 | 6 | 0
Not completed — Lost to Follow-up | 6 | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care | Total
Number analyzed (Participants) | 81 | 84 | 87 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 81 | 84 | 87 | 252
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.47 (3.13) | 7.37 (3.1) | 7.26 (3.02) | 7.37 (3.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 39 | 34 | 98
  Male | 56 | 45 | 53 | 154
Region of Enrollment [Number; unit: participants]
  United States | 81 | 84 | 87 | 252

OUTCOME MEASURES:

1. Primary Outcome: Parent Proxy-Reported Health-related Quality of Life (Pediatric Quality of Life Inventory)
Description: The PedsQL™ 4.0 Generic Core Scales Total Scale Score (PedsQL™), which has been shown to be internally consistent, valid, and responsive to indicators of clinical change for children with asthma (Chan, Mangione-Smith, Burwinkle, Rosen, & Varni, 2005; Seid et al., in press; Varni et al., 2004). The 23-item PedsQL™ asks respondents how often various issues have been a 'problem' in the past month, yields a score of 0 to 100 (higher scores are better), and includes parallel child self-report (ages 5-18 years) and parent proxy-report (ages 2-18 years) forms. We measured both self- and proxy-report, although our a priori primary outcome was parent proxy-report.
Time Frame: Baseline (T1), Post Intervention (3mo, T2), 6-month follow up (9mo post baseline, T3)
Population: All analyses were intent-to-treat and carried out according to a pre-established plan using SAS 9.1.3. All subjects with data at T2 or T3 were included in the analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care
Number analyzed (Participants) | 72 | 65 | 74
units on a scale | 81.2 (1.4) | 85.4 (1.5) | 80.8 (1.5)
Statistical Analysis 1: Comparison: Care Coordination+Problem Solving vs Standard Care; The primary effects of interest, condition and condition by time are fixed effects. PedsQL™ scores were analyzed as continuous normal outcomes with mixed effects regression models, which accounts for repeated measures over time for T2 and T3. Independent variables included baseline measure, time, asthma severity, condition, and condition by time interaction. We report the differences across groups in the adjusted mean changes over time; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — Bonferroni adjustment; Adjusted for child's age, race/ethnicity, Spanish, mother's education; Mean Difference (Net) = 4.0, 95% CI 2-sided [0.63 to 7.4]
Statistical Analysis 2: Comparison: Care Coordination vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — Bonferroni adjustment; Adjusted for child's age, race/ethnicity, Spanish, mother's education; Mean Difference (Net) = 3.1, 95% CI 2-sided [-0.21 to 6.4]

2. Secondary Outcome: Counts of Patients With One or More Asthma-related Emergency Department Visits.
Description: Utilization was measured by parent recall of emergency room visits for asthma over the last 6 months (at T1), 3 months (at T2), and 6 months (at T3).
Time Frame: Baseline (T1), Post Intervention (3mo, T2), 6-month follow up (9mo post baseline, T3)
Population: All analyses were intent-to-treat and carried out according to a pre-established plan using SAS 9.1.3.
Measure: Number; unit: participants
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care
Number analyzed (Participants) | 72 | 65 | 74
participants | 10 | 4 | 10
Statistical Analysis 1: Comparison: Care Coordination+Problem Solving vs Standard Care; Test type: Superiority or Other; p = 0.21, Regression, Logistic; Adjustment for age, race/ethnicity, Spanish language and mother's education; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.18 to 1.38]
Statistical Analysis 2: Comparison: Care Coordination vs Standard Care; Test type: Superiority or Other; p = 0.85, Regression, Logistic — adjustment for age, race/ethnicity, Spanish language and mother's education; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.53 to 2.83]

3. Secondary Outcome: Asthma Symptoms
Description: Asthma symptom frequency was measured via the number of days and nights with asthma symptoms over the past two weeks. Night time asthma symptoms were converted to number of subjects experiencing night time asthma symptoms more than 1 time per week.
Time Frame: Baseline (T1), Post Intervention (3mo, T2), 6-month follow up (9mo post baseline, T3)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care
Number analyzed (Participants) | 72 | 65 | 74
participants | 21 | 9 | 24
Statistical Analysis 1: Comparison: Care Coordination+Problem Solving vs Standard Care; Symptom frequency and utilization were analyzed using generalized linear mixed models (GLMM), with appropriate distribution and link functions. Nighttime symptoms is a dichotomous outcome and a logistic model was constructed; Test type: Superiority or Other; p = 0.011, Regression, Logistic; All analyses accounted for repeated measures and included the same terms in the model described previously; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.13 to 0.82]

ADVERSE EVENTS:
Arm/Group | Care Coordination | Care Coordination+Problem Solving | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/84 | 0/87
Other Adverse Events (participants affected / at risk) | 0/81 | 0/84 | 0/87

LIMITATIONS AND CAVEATS:
Substantial dropout, particularly from CC+PST, is a limitation. Our sample size was not large enough, nor was there sufficient variability in our secondary outcomes, to detect differences in health care utilization despite the odds ratios.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No